CLINICAL TRIAL: NCT05786287
Title: Long-term Safety of Umbilical Cord-Mesenchymal Stem Cell (UC-MSC) Transplantation in Patients With Retinitis Pigmentosa
Brief Title: Long-term Safety of UC-MSC Transplantation in Patients With Retinitis Pigmentosa
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Sponsor
Other Study IDs: CT/RP/08/2022
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Retinitis Pigmentosa
Keywords: Allogeneic Mesenchymal Stem Cell; Umbilical Cord Mesenchymal Stem Cell; Conditioned Medium; Allogeneic Umbilical Cord Mesenchymal Stem Cell; Safety
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Culture Media, Conditioned

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conditioned Medium (CM): 2 ml volume of Conditioned Medium derived Umbilical Cord Mesenchymal Stem Cell injected into peribulbar
  Interventions: Biological: Conditioned Medium (CM)
- UC-MSC + NaCl: 1.8 ml cell preparations are suspended in physiological NaCl until it reaches a 2 ml volume of cell suspension. Umbilical Cord Mesenchymal Stem Cell (UC-MSC) suspension injected into peribulbar
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cell (UC-MSC)
- UC-MSC+CM: 1.8 ml cell preparations are suspended in Conditioned Medium (CM) until it reaches a total of 2 ml volume of cell suspension. Umbilical Cord Mesenchymal Stem Cell (UC-MSC) + Conditioned Medium (CM) suspension injected into peribulbar
  Interventions: Biological: Conditioned Medium (CM); Biological: Umbilical Cord Mesenchymal Stem Cell (UC-MSC)

INTERVENTIONS:
Biological: Conditioned Medium (CM) — Conditioned Medium (CM) injected by peribulbar
  Groups: Conditioned Medium (CM); UC-MSC+CM
Biological: Umbilical Cord Mesenchymal Stem Cell (UC-MSC) — Umbilical Cord Mesenchymal Stem Cell (UC-MSC) injected by peribulbar
  Groups: UC-MSC + NaCl; UC-MSC+CM

SUMMARY:
The study will perform to follow-up UC-MSCs and CM transplantation. 18 patients will be called back to be examined after 5 years of UC-MSC and/or CM transplantation.

DETAILED DESCRIPTION:
The study will be performed on 18 patients who received UC-MSC and CM transplantation in 2018. The study is included as retrospective cohort since the transplantation happened 5 years ago. Patients will do a visual field test, visual acuity test, electroretinography, funduscopy, and Optical Coherence Tomography examination. The observation results will be written in the observation table and analyzed by a statistic.The study will be performed at Rumah Sakit Jakarta Eye Center and Rumah Sakit Umum Pusat Dr. Sardjito Yogyakarta.

ELIGIBILITY:
Inclusion Criteria:

* Visual field defects at the initial examination with Humphrey perimetry are between 25% to 50%
* Willing to sign informed consent as research subjects
* Willing to do the peribulbar injection with mesenchymal stem cells isolated from umbilical cord tissue
* Willing to do visual field checks with Humphrey's perimetry, vision tests with Snellen boards, Optical Coherent Tomography (OCT) examinations, electroretinogram examinations and fill out a quality of life questionnaire

Exclusion Criteria:

* Pregnant or nursing women
* Positive result of HIV test
* Have a history of eye tumours
* In the immunosuppressive treatment or other drugs that can affect the growth of transplanted stem cells
* Have another eye disease such as diabetic retinopathy, uveitis, cataract, and glaucoma
* Do not come to control according to the schedule determined by the researcher (loss to follow up)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retinitis Pigmentosa patients who have been transplanted UC-MSC and/or CM 5 years ago under clinical trials NCT04315025
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-13 (Estimated); Study Completion 2025-07-13 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity Test | 5 years after injection
  a test to see the sharpness of vision using Snellen Chart which is read at a distance of 6 meters. Normal eye test results are stated in 6/6.
Visual Field Test | 5 years after injection
  a test to assess the breadth of views of the lateral, medial, superior and inferior aspects using Humprey's perimetry.
Funduscopy | 5 yeas after injection
  an examination to see and assess the abnormalities and conditions in the ocular fundus using an ophthalmoscope. This examination is carried out by an ophthalmologist.
Electrorectinography | 5 years after injection
  an examination to provide a picture of objectivity, a quantitative measure of retinal function to monitor the function of stem cells and ganglion cells in the eye. This examination is carried out by a trained ophthalmologist.
Optical Coherence Tomography (OCT) | 5 years after injection
  is a diagnostic test that give the information about posterior segment structure, which is retina and optic nerve papillae so that it can be used to assess macular abnormalities
Angiography | 5 years after injection
  a process of taking photos of the retina by injecting fluorescent to get a bleeding location on the retina.

CONTACTS AND LOCATIONS:
Overall Officials: dr. Muhammad B Sasongko, Sp.M, M.Epid, PhD, Principal Investigator — Gadjah Mada University, Faculty of Medicine; dr Cosmos O Mangunsong, Sp.M, Study Director — Jakarta Eye Center; dr. Rifa Widyaningrum, M.Sc, PhD, Study Chair — Sardjito Hospital; Rima Haifa, S.Si, Study Chair — Prodia StemCell Indonesia; Marsya N Kirana, S.T., M.Sc, Study Chair — Prodia StemCell Indonesia
Locations (2):
- Indonesia (2):
  - Jakarta Eye Center Hospital, Jakarta, DKI Jakarta
  - Sardjito Hospital, Yogyakarta, Special Region